CLINICAL TRIAL: NCT03798444
Title: An Observational and Cross-sectional Study on Prevalence of Vertebral Fractures in Postmenopausal Women Living in Chinese Communities
Brief Title: Height Loss, Kyphosis Indicators, Bone Mineral Density and Vertebral Fractures in Chinese Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, ChenRong, Principal Investigator, Central South University
Other Study IDs: CRong
Record Dates: First submitted 2018-11-20; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Osteoporosis Fracture
Keywords: Height loss, Kyphosis; Osteoporosis, Vertebral fracture; Postmenopausal women
MeSH Terms: conditions — Osteoporotic Fractures; Kyphosis; Osteoporosis; Spinal Fractures | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone mineral denstiy: BMD of the lumbar spine, left femoral neck, and total hip were measured using dual energy X-ray absorptiometry in all subjects.Accroding to The World Health Organization, we defined osteoporosis as a T-score ≤-2.5,and the non osteoporosis as T-score>-2.5.
  Interventions: Radiation: dual energy X-ray absorptiometry
- Vertebral fractures: VFs were assessed using lateral spine imaging from T4 to L4 on X-ray. A visual semi-quantitative method was used, with fractures defined as a vertebral height ratio <0.80 for the anterior/posterior or middle/posterior height ratio within a vertebra, or the posterior/posterior height ratio when compared to an adjacent vertebra.
  Interventions: Radiation: lateral spine imaging from T4 to L4 on X-ray

INTERVENTIONS:
Radiation: dual energy X-ray absorptiometry — BMD of the lumbar spine, left femoral neck, and total hip were measured using dual energy X-ray absorptiometry. The lumbar spine, left femoral neck, or total hip of T-score ≤-2.5 as the osteoporosis
  Groups: Bone mineral denstiy
Radiation: lateral spine imaging from T4 to L4 on X-ray — VFs were assessed using lateral spine imaging from T4 to L4 on X-ray .A visual semi-quantitative method was used, with fractures defined as a vertebral Vertebral fractures should be diagnose if height ratio <0.80 for the anterior/posterior or middle/posterior height ratio within a vertebra, or the posterior/posterior height ratio when compared to an adjacent vertebra
  Groups: Vertebral fractures

SUMMARY:
This is an observational and cross-sectional study on the height loss, kyphosis indicators, bone mineral density and vertebral fractures in Chinese postmenopausal women

DETAILED DESCRIPTION:
Postmenopausal women (N=255) aged ≥50 years were randomly selected from community centers in Changsha City, Hunan Province, China in September 2017. Menopause was defined as the absence of menstrual cycles for at least one year. All subjects were noninstitutionalized and in good health.The criteria for exclusion were morphological abnormalities or skeletal distortions that prohibited either clinical measurements or morphometric assessments of skeletal radiographs All participants were interviewed using a standard questionnaire. Body weight and height were measured to the closest 0.1 kg and 0.5 cm, respectively, with subjects wearing light clothing and no shoes. Current height was measured using a wall-mounted stadiometer, with a horizontal plate pressed on the head, and hair flattened. All subjects provided basic information, including current age, age at the start of menopause, years since menopause (YSM), weight, and their tallest recalled height. The current measured height subtracted from the tallest recalled height was subjects' HHL.The RPD, which was the vertical distance between the lowest margin of the ribs and the superior surface of the iliac crest along the mid-axillary line, was measured twice by a physician who stood behind the subject. For the kyphosis assessment, subjects were measured without shoes, with their heels, buttocks, and back to the wall, and head in a horizontal position with a double chin shown. The wall-occiput distance was defined as the horizontal distance between the wall and the back of the head. The distance between the prominence of the 7th cervical vertebra and the wall was defined as 7th cervical vertebra-wall distance (C7WD) , and wall-tragus-distance (WTD) was defined as the horizontal distance from the participant's tragus to the wall . All RPD and anthropometric indicators of kyphosis were measured in increments of 0.1 cm by two trained physicians.BMD of the lumbar spine, left femoral neck, and total hip were measured using dual energy X-ray absorptiometry. VFs were assessed using lateral spine imaging from T4 to L4 on X-ray.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women aged ≥50 years (Menopause was defined as the absence of menstrual cycles for at least one year)

Exclusion Criteria:

Morphological abnormalities or skeletal distortions

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged ≥50 years were randomly selected from community centers in Changsha City, Hunan Province, China in September 2017.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Height | 4 weeks
  Subjects wearing light clothing and no shoes. Current height was measured using a wall-mounted stadiometer, with a horizontal plate pressed on the head, and hair flattened. Height were measured to the closest 0.5 cm,
Weight | 4 weeks
  Body weight was measured with subjects wearing light clothing and no shoes
Rib to pelvis distance | 4 weeks
  The rib to pelvis distance, which was the vertical distance between the lowest margin of the ribs and the superior surface of the iliac crest along the mid-axillary line, was measured twice by a physician who stood behind the subject. Measured in increments of 0.1 cm by two trained physicians.
Wall-occiput distance | 4 weeks
  Subjects were measured without shoes, with their heels, buttocks, and back to the wall, and head in a horizontal position with a double chin shown. The wall-occiput distance was defined as the horizontal distance between the wall and the back of the head. Measured in increments of 0.1 cm by two trained physicians.
7th cervical vertebra-wall distance | 4 weeks
  Subjects were measured without shoes, with their heels, buttocks, and back to the wall, and head in a horizontal position with a double chin shown. The distance between the prominence of the 7th cervical vertebra and the wall was defined as 7th cervical vertebra-wall distance. Measured in increments of 0.1 cm by two trained physicians.
Wall-tragus-distance | 4 weeks
  Subjects were measured without shoes, with their heels, buttocks, and back to the wall, and head in a horizontal position with a double chin shown.Wall-tragus-distance was defined as the horizontal distance from the participant's tragus to the wall. Measured in increments of 0.1 cm by two trained physicians.
Historical height loss | 4 weeks
  The current measured height subtracted from the tallest recalled height was subjects' historical height loss

CONTACTS AND LOCATIONS:
Overall Officials: sheng zhifeng, MD, Principal Investigator — Central south of university
Locations (1):
- The 2nd Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoh K, Kuwabara A, Tanaka K. Detective value of historical height loss and current height/knee height ratio for prevalent vertebral fracture in Japanese postmenopausal women. J Bone Miner Metab. 2014 Sep;32(5):533-8. doi: 10.1007/s00774-013-0525-y. PMID 24122280
- [Background] Siminoski K, Warshawski RS, Jen H, Lee K. The accuracy of historical height loss for the detection of vertebral fractures in postmenopausal women. Osteoporos Int. 2006 Feb;17(2):290-6. doi: 10.1007/s00198-005-2017-y. Epub 2005 Sep 6. PMID 16143833
- [Background] Siminoski K, Warshawski RS, Jen H, Lee KC. Accuracy of physical examination using the rib-pelvis distance for detection of lumbar vertebral fractures. Am J Med. 2003 Aug 15;115(3):233-6. doi: 10.1016/s0002-9343(03)00299-7. No abstract available. PMID 12935830
- [Background] Mizukami S, Abe Y, Tsujimoto R, Arima K, Kanagae M, Chiba G, Aoyagi K. Accuracy of spinal curvature assessed by a computer-assisted device and anthropometric indicators in discriminating vertebral fractures among individuals with back pain. Osteoporos Int. 2014 Jun;25(6):1727-34. doi: 10.1007/s00198-014-2680-y. Epub 2014 Mar 14. PMID 24627138
- [Background] Suwannarat P, Amatachaya P, Sooknuan T, Tochaeng P, Kramkrathok K, Thaweewannakij T, Manimmanakorn N, Amatachaya S. Hyperkyphotic measures using distance from the wall: validity, reliability, and distance from the wall to indicate the risk for thoracic hyperkyphosis and vertebral fracture. Arch Osteoporos. 2018 Mar 12;13(1):25. doi: 10.1007/s11657-018-0433-9. PMID 29532182
- [Background] Ralston SH, Urquhart GD, Brzeski M, Sturrock RD. Prevalence of vertebral compression fractures due to osteoporosis in ankylosing spondylitis. BMJ. 1990 Mar 3;300(6724):563-5. doi: 10.1136/bmj.300.6724.563. PMID 2108749

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT03798444/Prot_SAP_000.pdf